CLINICAL TRIAL: NCT04784845
Title: Lactamica 9: Defining Upper Respiratory Colonisation and Microbiome Evolution in Mother-infant Pairs Following Neisseria Lactamica Inoculation in Late Pregnancy
Brief Title: Lactamica 9: Neisseria Lactamica Inoculation in Late Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University of Edinburgh (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 61640
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Microbial Colonization
Keywords: Human challenge study; Controlled human infection; Neonatal microbiome; Pregnancy; Respiratory Tract Infections; Meningitis; Respiratory microbiome
MeSH Terms: conditions — Communicable Diseases; Respiratory Tract Infections; Meningitis

STUDY DESIGN:
Intervention Model Description: A single intervention cohort will receive one open label intervention (nasal inoculation with 10^5 CFU N. lactamica).
  If any naturally-occurring N. lactamica carriers are identified at screening, they will not attend for inoculation with N. lactamica, but will be invited to remain in the study. They (and their neonates) will undergo the same follow-up visits and sampling as inoculated volunteers. This observational cohort is not considered a separate study arm, and there is no recruitment target for this cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N. lactamica Y92-1009 (Experimental): Nasal inoculation with 10^5 CFU N. lactamica in 1ml phosphate-buffered saline via pipette to both nostrils; single inoculation at 36+0 to 37+6 weeks gestation
  Interventions: Biological: N. lactamica Y92-1009

INTERVENTIONS:
Biological: N. lactamica Y92-1009 — Lyophilised N. lactamica reconstituted in phosphate-buffered saline

SUMMARY:
Bacteria living in the nose and throat are generally harmless, but in some circumstances cause infections of the lungs (pneumonia) and brain (meningitis), which are among the commonest causes of death worldwide in young children (especially newborns). Babies with certain 'good' bacteria in the nose and throat are less likely to have infections by such 'bad' bacteria. Scientists have tried giving probiotics ('good' bacteria swallowed or sprayed into the nose) to pregnant women, new mothers and babies. These studies show that many probiotics are safe, but the amount of bacteria given is often unknown, and it is unclear if they work. A more precise option is to use controlled inoculation, by inserting a specific amount of particular 'good' bacteria into the nose under carefully controlled conditions. Our team have previously shown that inoculation with Neisseria lactamica ('good' bacteria) safely and reliably decreases Neisseria meningitidis ('bad' bacteria) in healthy adults' noses. N. lactamica is a type of harmless bacteria found in over 40% of children aged 1-2 years, but is uncommon in newborns and adults.

We plan to inoculate 20 healthy pregnant women with N. lactamica nose drops, to find out if it is transferred to their babies after birth. Newborns become rapidly covered (colonised) with bacteria from their mothers, other people, and the environment, so this method mimics a natural way that babies receive bacteria. We will take saliva and nose swabs one day, one week, one month and four months after birth, and will use microbiological and genetic methods to study how the bacteria changes in babies compared with their mothers.

DETAILED DESCRIPTION:
We plan to perform nasal inoculation with N. lactamica (wild type strain Y92-1009) in healthy pregnant women, to establish whether horizontal N. lactamica transfer to their neonates occurs, and to characterise the impact on the developing neonatal upper respiratory tract (URT) microbiome. If successful, this study will provide a novel model for inducing and capturing a natural colonisation event in neonates. Unlike traditional controlled human infection models, which capture inoculation-induced colonisation, this first-in-man model would study person-to-person commensal transmission, allowing comparison of microbiome changes and adaptive commensal microevolution in mother-infant pairs. We have already conducted relevant Patient and Public Involvement research, in which all 12 pregnant women interviewed reported approval for this proposed study, and 11 expressed that they would have been interested in taking part in such a study.

We will approach healthy pregnant women in their second and third trimesters of pregnancy. Eligibility screening and enrolment will take place at 34+0 to 36+6 weeks gestation, and 20 women (not already colonised with N. lactamica) will be inoculated nasally with 10^5 colony forming units N. lactamica Y92-1009 at 36+0 to 37+6 weeks gestation. Samples will be obtained from new mothers (nasopharyngeal, oropharyngeal and saliva) and their neonates (nasopharyngeal and saliva) at 1 day, 1 week, 1 month and 4 months post-partum. If possible, and with the volunteer's consent, we will collect an umbilical cord blood sample at delivery and an infant venous blood sample at 1 month and 4 months post-partum, for storage and use in future studies. We will also collect a maternal venous blood sample at 4 months post-partum, as well as a saliva swab from any household contacts aged under 5 years. Any natural N. lactamica carriers identified at screening will not be inoculated, but will be followed-up with their neonates for biological sampling.

Pharyngeal and saliva swabs will be suspended in storage medium, aliquoted and stored at -80°C. N. lactamica colonisation will be confirmed using selective agar, Gram stain, microscopy, and analytical profile index testing (and matrix-assisted laser desorption/ionization time-of-flight for inconclusive results). N. lactamica colonisation density will be quantified, isolates will be stored at -80°C, and Y92-1009 strain identity will be confirmed using targeted polymerase chain reaction (PCR).

Microbiome analysis will be performed on thawed aliquots of paired mother-neonate samples, by DNA extraction, 16S ribosomal ribonucleic acid (rRNA) gene PCR, and amplicon sequencing. Poor quality and chimeric sequence reads will be removed, and high quality reads will be trimmed, aligned and clustered for taxonomic classification and statistical analysis.

Paired maternal and neonatal isolates confirmed as N. lactamica Y92-1009 will be sequenced, and resulting genomes will be mapped to a complete N. lactamica Y92-1009 closed reference genome, to assess for evidence of distinct microevolution.

We will also compare paired microbiome profiles to identify candidate organisms that are present in mothers and their infants. Paired mother-neonate sample aliquots will be thawed and plated onto selective media, and isolates of candidate species will be identified using Gram stain, microscopy, and other relevant microbiological tests. Resulting isolates will be sequenced and analysed for evidence of strain sharing between mothers and their neonates, suggesting horizontal transfer.

ELIGIBILITY:
Inclusion Criteria:

All the following inclusion criteria must apply in order for the volunteer to be eligible for the study:

* Healthy adult aged 18 years or over on the day of enrolment.
* Singleton pregnancy, 34+0 to 36+6 weeks gestation on the day of enrolment.
* Documentation of a 20-week ultrasound scan with no life-limiting congenital anomalies, and no maxillofacial / otorhinolaryngological / neuroanatomical anomalies.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Able and willing to give written informed consent to participate in the study.
* Booked to receive antenatal care at University Hospital Southampton NHS Foundation Trust.

Exclusion Criteria:

The volunteer may not enter the study if any of the following exclusion criteria apply:

* Any confirmed or suspected immunosuppressive or immunocompromised state, including: HIV infection; asplenia; recurrent severe infections; or use of immunosuppressant medication (for more than 14 days within the past 6 months, excluding topical and inhaled steroids).
* Planned use of immunosuppressant medication in later pregnancy or post-partum.
* Occupational, household or intimate contact with any immunosuppressed persons.
* Participation within the last 12 weeks in a clinical trial involving receipt of an investigational product, or planned use of an investigational product during the study period.
* Prior participation at any time in research studies involving inoculation with N. lactamica.
* Use of oral or intravenous antibiotics within 30 days prior to the N. lactamica inoculation visit.
* Planned use of oral or intravenous antibiotics at any time during the study period (e.g. for planned elective caesarean section or group B streptococcus colonisation).
* Allergy to soya or yeast.
* Previous stillbirth or neonatal death.
* Pre-pregnancy diabetes mellitus.
* Any other finding that may (in the Investigator's opinion): increase the risk to the volunteer (or their fetus/infant or close contacts) of participating in the study; affect the volunteer's ability to participate in the study and complete follow-up; or impair interpretation of study data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only healthy pregnant women will be recruited. Neonates of any gender will be included.
Enrollment: 31 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Neonatal N. lactamica colonisation | Up to 4 weeks post-partum
  Confirmation of neonatal (aged 0-30 days) N. lactamica colonisation by selective culture of biological (nasopharyngeal and/or saliva) samples

SECONDARY OUTCOMES:
Adverse reactions or serious adverse events | Enrolment (34+0 to 36+6 weeks gestation) to 4 weeks post-partum
  Percentage of participants (women and their neonates) with adverse reactions or serious adverse events within the study period
Neonatal N. lactamica Y92-1009 colonisation | Birth (0-24 hours post-partum), 7+/-3 days post-partum, 28+/-3 days post-partum
  Confirmation of N. lactamica Y92-1009 strain identity by targeted polymerase chain reaction in neonates found to be colonised with N. lactamica
N. lactamica colonisation kinetics | Birth (0-24 hours post-partum), 7+/-3 days post-partum, 28+/-3 days post-partum
  Characterisation of N. lactamica colonisation density in inoculated volunteers versus their infants across study time points and sample types
Upper respiratory microbiome | Birth (0-24 hours post-partum), 7+/-3 days post-partum, 28+/-3 days post-partum
  Characterisation of microbiome composition, alpha diversity (within one biological sample) and beta diversity (between different biological samples) in inoculated volunteers compared with their infants across study time points and sample types; and (if horizontal N. lactamica transfer is detected in at least some but not all infants) in infants colonised with N. lactamica compared with uncolonised infants.
N. lactamica Y92-1009 microevolution | Birth (0-24 hours post-partum), 7+/-3 days post-partum, 28+/-3 days post-partum
  If horizontal N. lactamica transfer is detected in at least some infants: N. lactamica genome sequence for isolates derived from inoculated volunteers compared with their infants across study time points and sample types, and comparison with an N. lactamica Y92-1009 closed reference genome

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Jones, Principal Investigator — University of Southampton; Robert C Read, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton NHS Foundation Trust, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Theodosiou AA, Bogaert D, Cleary DW, Dale AP, Gbesemete DF, Guy JM, Laver JR, Raud L, Jones CE, Read RC. Controlled human infection model of Neisseria lactamica in late pregnancy investigating mother-to-infant transmission in the UK: a single-arm pilot trial. Lancet Microbe. 2025 Apr;6(4):100986. doi: 10.1016/j.lanmic.2024.100986. Epub 2025 Feb 19. PMID 39986292
- [Derived] Bevan JHJ, Theodosiou AA, Corner J, Dorey RB, Read RC, Jones CE. A Questionnaire-based Study Exploring Participant Perspectives in a Perinatal Human Challenge Trial. Pediatr Infect Dis J. 2023 Nov 1;42(11):935-941. doi: 10.1097/INF.0000000000004036. Epub 2023 Jul 18. PMID 37463362
- [Derived] Theodosiou AA, Laver JR, Dale AP, Cleary DW, Jones CE, Read RC. Controlled human infection with Neisseria lactamica in late pregnancy to measure horizontal transmission and microbiome changes in mother-neonate pairs: a single-arm interventional pilot study protocol. BMJ Open. 2022 May 18;12(5):e056081. doi: 10.1136/bmjopen-2021-056081. PMID 35584870